CLINICAL TRIAL: NCT06324669
Title: Investigating the Blood Glucose Lowering Effect of Exogenous Ketone Ingestion in People With Type 2 Diabetes
Brief Title: The Effect of a Ketone Drink on Blood Glucose Levels in People With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University of British Columbia (Other); Medical Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 4765060
Record Dates: First submitted 2024-03-12; First posted 2024-03-22 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Randomised cross over trial counterbalanced for trial order
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Coded, known only to independent individual
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone supplementation (Experimental): 100 mL flavoured drink containing 0.3 g/kg ketone monoester ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate; ΔG®, University of Oxford; https://www.deltagketones.com)
  Interventions: Dietary Supplement: Ketone supplement
- Placebo (Placebo Comparator): Placebo with stevia and bitter agent to flavour match
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Ketone supplement — 100 mL flavoured drink containing 0.3 g/kg ketone monoester ((R)-3-hydroxybutyl (R)-3-hydroxybutyrate; ΔG®, University of Oxford; https://www.deltagketones.com) consumed 30 min prior to a mixed meal tolerance test, on 2 occasions during test day
  Arms: Ketone supplementation
Dietary Supplement: Placebo supplement — Placebo with stevia and bitter agent to flavour match, consumed 30 min prior to a mixed meal tolerance test, on 2 occasions during test day
  Arms: Placebo

SUMMARY:
Ketones are naturally produced by our body and can affect our blood sugar levels. Ketones could be important in the treatment of type 2 diabetes (T2D). The purpose of this research is to determine if a ketone drink can lower blood sugar in people with T2D following a meal. This research will provide new knowledge about the regulation of blood sugar. This may also inform if ketone drinks could be used as a treatment for T2D.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 41-70 years old
2. Body mass index 27-40 mg/m²
3. Type 2 diagnosis for more than 1 year
4. HbA1c >6%

Exclusion Criteria:

1. Currently following ketogenic diet
2. Use of insulin
3. HbA1c >10%
4. Recent weight loss (>5kg in 6 months)
5. Recent eGFR <30mL/min
6. Heart failure
7. Substance abuse
8. Cancer
9. Myocardial infarction within 6 months
10. Pregnancy or consideration of
11. Use of antipsychotic drugs

Ages: 41 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-03-16 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
Rate of endogenous glucose production | 4 hours
  Rate of endogenous glucose production over 4 hours in response to a meal measured by blood sample

SECONDARY OUTCOMES:
Total rate of glucose appearance | 4 and 8 hours
  Total rate of glucose appearance measured using the change in glucose enrichment/concentration over 4 and 8 hours following a meal
Exogenous glucose rate of appearance | 4 and 8 hours
  Exogenous rate of glucose appearance measured using the change in glucose enrichment/concentration over 4 and 8 hours following a meal
Total rate of glucose disappearance | 4 and 8 hours
  Total rate of glucose disappearance measured using the change in glucose enrichment/concentration over 4 and 8 hours following a meal
Rate of gluconeogenesis | 4 and 8 hours
  Rate of gluconeogenesis measured using the change in glucose enrichment/concentration over 4 and 8 hours following a meal
Rate of glycogenolysis | 4 and 8 hours
  Rate of glycogenolysis measured using the change in glucose enrichment/concentration over 4 and 8 hours following a meal
Beta-cell function | 4 and 8 hours
  Beta-cell function using dynamic modelling of insulin/c-peptide secretion over 4 and 8 hours following a meal
Insulin concentration | 4 and 8 hours
  Insulin concentration using ELISA assay over 4 and 8 hours following a meal
Glucagon concentration | 4 and 8 hours
  Glucagon concentration using ELISA assay over 4 and 8 hours following a meal
GLP-1 concentration | 4 and 8 hours
  GLP-1 using ELISA assay over 4 and 8 hours following a meal
GIP concentration | 4 and 8 hours
  GIP concentration using ELISA assay over 4 and 8 hours following a meal
Glycerol concentration | 4 and 8 hours
  Glycerol concentration using colorimetric assay over 4 and 8 hours following a meal
Free fatty acid concentration | 4 and 8 hours
  Free fatty acids using colorimetric assay over 4 and 8 hours following a meal
Ketone concentration | 4 and 8 hours
  Ketone concentration using colorimetric assay over 4 and 8 hours following a meal
Energy expenditure | 4 and 8 hours
  Energy expenditure using indirect calorimetry over 4 and 8 hours following a meal

CONTACTS AND LOCATIONS:
Overall Officials: Francis B Stephens, PhD, Principal Investigator — University of Exeter
Locations (1):
- Sport & Health Sciences University of Exeter, Exeter, Devon, United Kingdom